CLINICAL TRIAL: NCT05763615
Title: 3D Modeling of the Cervico-facial Region and Cranial Nerve Tractography: IMAG 2 ORL Project
Acronym: IMAG 2 ORL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP230015; 2020-A02279-30 (Other: ID-RCB Number)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Neoplasms; Congenital Abnormalities
Keywords: 3D modeling of the cervico-facial region; Tractography MRI; Diffusion tensor magnetic resonance imaging (DT-MRI); Cranial nerve; Pediatrics
MeSH Terms: conditions — Head and Neck Neoplasms; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Children aged 1 to 5 benefiting from a 3T MRI at the Necker Enfants-Malades hospital as part of the initial assessment of a tumor or cervico-facial malformation and at the first postoperative follow-up MRI if indicated for the care during a period of 12 months.
  Interventions: Other: Tractography MRI
- Control patients (Experimental): Children aged 1 to 5 benefiting from a 3T MRI at the Necker Enfants-Malades hospital as part of the initial assessment of an ENT pathology other than that of the patient group.
  Interventions: Other: Tractography MRI

INTERVENTIONS:
Other: Tractography MRI — Addition to the sequences usually done for the care of these patients (CubeT2, Diffusion, CubeT1, CubeT2 fiesta, ASL, T1 injected with gadolinium), of a so-called "research" tractography sequence benefiting from CE marking and not requiring specific injection.
  Search sequence acquisition time: 10 minutes.

SUMMARY:
3D modeling associated with the tracking of nerve fibers meets the needs of preoperative planning for tumors and cervico-facial congenital malformations. Indeed, these lesions are closely related to the cranial nerves and in particular nerve V (infratemporal fossa), nerve VII (temporal bone, parotido-masseter region), nerves IX, X, XI, XII and the chain cervical sympathetic (infratemporal and cervical regions). The development of a model of this region will therefore improve the surgical management of these children.

DETAILED DESCRIPTION:
Children aged 1 to 5 benefiting from a 3T magnetic resonance imaging (MRI) at the Necker Enfants-Malades hospital for their care, meeting the inclusion criteria and participating in the study, will benefit during their MRI from the care, a sequence "Research" tractography MRI lasting 10 minutes. This sequence is already validated and proposed for tractography but in specialties other than pediatric ENT.

Tractography techniques are mathematical algorithms based on the diffusion tensor (micro-movements of water molecules in tissues) to reconstruct the path of nerve fibers in each volume unit of the MRI image (voxel).

3D modeling associated with the tracking of nerve fibers meets the needs of preoperative planning for tumors and cervico-facial congenital malformations. Indeed, these lesions are closely related to the cranial nerves.

ELIGIBILITY:
Inclusion Criteria:

* Benefiting from social security scheme.
* Informed consent signed by holders of parental authority and the investigator.
* Patient group: children aged 1 to 5 benefiting from a 3T MRI at the Necker Enfants-Malades hospital as part of the initial assessment of a tumor or a cervico-facial malformation.
* Control group: children aged 1 to 5 benefiting from a 3T MRI at the Necker Enfants-Malades hospital as part of the initial assessment of an ENT pathology other than that of the patient group (examples: velar insufficiency, congenital deafness).

Exclusion Criteria:

Child with a contraindication to MRI: allergy to contrast product, pacemaker, Starr Edwards valves, stent placed for less than 6 weeks, vascular clips, contraindication to sedation.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
Implementation of a tractography algorithm | 24 months
  Imagery analysis of tractography MRI and implementation of a tractography algorithm.

SECONDARY OUTCOMES:
Evaluate the correlation between the 3D modeling and the intraoperative findings | At the operation
  Evaluate the correlation between the 3D modeling and the intraoperative findings. Intraoperative evaluation of the position of the facial nerve and its relationship to the tumor.
Course of the cranial nerves in children | 24 months
  Compare the course of the cranial nerves in children treated for tumor or congenital malformation compared to control patients treated for another ENT pathology: comparison of images obtained between patients and controls (radiological analysis).
Assess the presence of post-treatment sequelae nerve lesions | 12 months
  Assess the presence of post-treatment sequelae nerve lesions for subject patients (surgery or radiochemotherapy) on follow-up MRI: during follow-up MRIs, analysis by tractography of the nerve related to the lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Romain Luscan, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basser PJ, Pajevic S, Pierpaoli C, Duda J, Aldroubi A. In vivo fiber tractography using DT-MRI data. Magn Reson Med. 2000 Oct;44(4):625-32. doi: 10.1002/1522-2594(200010)44:43.0.co;2-o. PMID 11025519
- [Background] Beaulieu C. The basis of anisotropic water diffusion in the nervous system - a technical review. NMR Biomed. 2002 Nov-Dec;15(7-8):435-55. doi: 10.1002/nbm.782. PMID 12489094
- [Background] Jacquesson T, Frindel C, Kocevar G, Berhouma M, Jouanneau E, Attye A, Cotton F. Overcoming Challenges of Cranial Nerve Tractography: A Targeted Review. Neurosurgery. 2019 Feb 1;84(2):313-325. doi: 10.1093/neuros/nyy229. PMID 30010992
- [Background] Yoshino M, Abhinav K, Yeh FC, Panesar S, Fernandes D, Pathak S, Gardner PA, Fernandez-Miranda JC. Visualization of Cranial Nerves Using High-Definition Fiber Tractography. Neurosurgery. 2016 Jul;79(1):146-65. doi: 10.1227/NEU.0000000000001241. PMID 27070917
- [Background] Jacquesson T, Cotton F, Attye A, Zaouche S, Tringali S, Bosc J, Robinson P, Jouanneau E, Frindel C. Probabilistic Tractography to Predict the Position of Cranial Nerves Displaced by Skull Base Tumors: Value for Surgical Strategy Through a Case Series of 62 Patients. Neurosurgery. 2019 Jul 1;85(1):E125-E136. doi: 10.1093/neuros/nyy538. PMID 30476219
- [Background] Muller CO, Mille E, Virzi A, Marret J-B, Peyrot Q, Delmonte A, et al. Integrating tractography in pelvic surgery: a proof of concept. J Pediatr Surg Case Rep. 1 sept 2019;48:101268